CLINICAL TRIAL: NCT05928507
Title: CSP0010 FINDER® Instrument and FINDER® FLU A/B, RSV, SARS-CoV-2 Test Clinical Evaluation Protocol
Brief Title: FINDER® Instrument and FINDER® FLU A/B, RSV, SARS-CoV-2 Test Clinical Evaluation Protocol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Baebies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP0010
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Influenza A; Influenza Type B; SARS CoV 2 Infection; RSV Infection
MeSH Terms: conditions — COVID-19; Respiratory Syncytial Virus Infections | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Adult Category 1 -fresh prospective: NP swabs from the Adult population >17 years, collected prospectively from adults presenting with symptoms of respiratory illness. Tested within 72 hours of collection.
  Interventions: Diagnostic Test: Diagnostic Test for identification of influenzas A, influenzas B, RSV and SARS-CoV-2 infections
- Pediatric Category 1 -fresh prospective: P swabs from the pediatric population <=17 years, collected prospectively from pediatrics presenting with symptoms of respiratory illness. Tested within 72 hours of collection.
  Interventions: Diagnostic Test: Diagnostic Test for identification of influenzas A, influenzas B, RSV and SARS-CoV-2 infections
- Adult Category 2 -frozen prospective: NP swabs from the Adult population >17 years, were collected prospectively from adults presenting with symptoms of respiratory illness. Frozen following CLSI guidelines to be Tested at a later time point approximately 3 months.
  Interventions: Diagnostic Test: Diagnostic Test for identification of influenzas A, influenzas B, RSV and SARS-CoV-2 infections
- Pediatric Category 2 -frozen prospective: NP swabs from the pediatric population >17 years, were collected prospectively from pediatrics presenting with symptoms of respiratory illness. Frozen following CLSI guidelines to be tested at a later time point approximately 3 months.
  Interventions: Diagnostic Test: Diagnostic Test for identification of influenzas A, influenzas B, RSV and SARS-CoV-2 infections

INTERVENTIONS:
Diagnostic Test: Diagnostic Test for identification of influenzas A, influenzas B, RSV and SARS-CoV-2 infections — The FINDER FLU A/B, RSV, SARS-CoV-2 Test real-time RT-PCR test for the qualitative detection of viral RNA from RSV, FLU A, FLU B and SARS-CoV-2 in nasopharyngeal (NP) specimens from individuals suspected of respiratory tract infection by their healthcare provider.
  Nucleic acids from respiratory viruses identified by this test are typically detectable in nasopharyngeal swabs (NP) during the acute phase of infection. The detection and identification of specific viral nucleic acids from individuals signs is an indication of the presence of the identified microorganism and assist in the diagnosis of respiratory infection when considered alongside other clinical and epidemiological information.

SUMMARY:
The goal of this observational study is to compare the FINDER FLU A/B, RSV, SARS-CoV-2 Test to an FDA-cleared device. The study will utilize prospectively collected de-identified nasopharyngeal samples obtained from both pediatric and adult populations from subjects presenting with symptoms of respiratory illness.

The main question it aims to answer are:

• the study is to validate that the device intended use in terms that the device's performance meets the criteria for substantial equivalence with a predicate and satisfies the statutory criteria for Clinical Laboratory Improvement Amendments (CLIA) waiver.

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal samples will be collected using swabs and placed in liquid transport media.
* The samples are obtained from individuals exhibiting respiratory signs and symptoms.
* These samples are collected as part of standard differential diagnostic procedures.
* A minimum sample volume of 1.5 mL is required for testing purposes.

Exclusion Criteria:

* de-identified samples that have not been stored in accordance with CDC recommendations for nasopharyngeal (NP) sample storage.
* Samples obtained from subjects who do not exhibit signs or symptoms of respiratory illness.
* The sample with a volume is less than 1.5 mL

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this protocol will consist of samples collected from adult and pediatric individuals with signs and symptoms of respiratory disorders.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative detection of viral RNA from Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), Influenza A (H1N1 and H3N2 subtypes), Influenza B (Victoria and Yamagata strains), and Respiratory Syncytial Virus (A and B subtypes) | within 72 hours of collection of NP swab
  Qualitative detection of viral RNA from Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), Influenza A (H1N1 and H3N2 subtypes), Influenza B (Victoria and Yamagata strains), and Respiratory Syncytial Virus (A and B subtypes) in nasopharyngeal (NP) specimens from individuals suspected of respiratory tract infection by their healthcare provider.for adults and pediatrics when compared to a known FDA cleared assay/ instrument combination.

SECONDARY OUTCOMES:
CLIA Waived results and clinical laboratory result | within 72 hours of collection of NP swab
  Characterization of the performance of the FINDER device when used at a CLIA-waived location and when used in a clinical laboratory location.

CONTACTS AND LOCATIONS:
Overall Officials: Candice Prowse, Study Director — Baebies, Inc.
Locations (1):
- Wake Med, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data. The data is in support of a 510K